CLINICAL TRIAL: NCT04095897
Title: Does Pecs II Block Reduce the Incidence of Post Mastectomy Pain Syndrome (PMPS)? A Cross Sectional Study
Acronym: PMPS
Status: Completed | Type: Observational
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Other Study IDs: FF-2018-084; NMRR ID: 17-2627-38056 (Registry Identifier: National Medical Research Register)
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Chronic Pain
Keywords: PMPS; Pecs II; Pectoral Nerve Block; CPSP
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- conventional analgesic therapy: Patient underwent mastectomy with conventional analgesic therapy
- Pecs II block: Patient underwent mastectomy with conventional analgesic therapy with pre induction Pecs II block
  Interventions: Procedure: Pecs II Block

INTERVENTIONS:
Procedure: Pecs II Block — Peripheral nerve block - Regional anesthesia : Pectoral Nerve block type 2
  Groups: Pecs II block

SUMMARY:
Post mastectomy pain syndrome (PMPS) is a chronic pain condition that develops after breast cancer surgery. The objective of this study was to determine if Pecs II block administered prior to general anesthesia (GA) reduced the incidence of PMPS after mastectomy and axillary clearance (MAC) when compared with conventional analgesic therapy.

DETAILED DESCRIPTION:
This cross sectional study was approved by the research and ethics committees in both institutional and national levels. This project was registered under National Medical Research Register (NMRR), Ministry of Health Malaysia.

Patients who underwent MAC from July 2015 - June 2017 in Hospital Kuala Lumpur (HKL) were recruited. In order to standardize surgical technique and reduce confounding factors, case selection was only limited to unilateral MAC. Other breast cancer surgeries, such as wide local excision, modified radical mastectomy (MRM) and lumpectomy, were excluded. Patients with the following characteristics and problems were excluded from our study - past history of chronic pain and on regular analgesics, chemotherapy or radiotherapy before surgery, surgical complications (such as infection or wound breakdown) or cancer recurrence, history of psychiatric illness, inability to be contacted, inability or unwillingness to participate in the study.

There is currently no standard definition for this chronic pain syndrome. Depending on the definitions applied, patient selection and methods used, the incidence varies. The definition of PMPS used in this study was modified from International Association for the Study of Pain19 (IASP) and other studies.9,20 In our study, PMPS is taken as chronic post surgical pain in the anterior aspect of the thorax, axilla, and/or upper half of the arm beginning after mastectomy, without objective evidence of local abnormality, persisting either continuously or intermittently for more than three months after surgery, and may be associated with allodynia or sensory loss.

Questionnaire used in this study was obtained with permission from Dr Manoj Kumar Karmakar, the author of a previous study on the effect of thoracic paravertebral block (TPVB) on chronic pain post mastectomy.21 It was prepared in both English and Malay versions (Appendix 1) to cater for our local population. The English version was translated to Malay using forward and retrograde translation methods to check the reliability and precision of the words by four independent translators who were bicultural Malay speakers with a good command of English. The translation was further evaluated by a panel of experts in the field of Regional Anesthesia and Pain Management to verify the idiomatic and cross-cultural equivalence to the English version. Seven respondents were then recruited to assess face validity of the questionnaire. Repeat evaluation was done until respondents understood all the questions in the process of content validation. No modification was needed as the first draft of questionnaire was well understood by all respondents. Internal consistency reliability and construct validation was done using Cronbach's alpha, Kaiser-Meyer-Olkin (KMO) test and Bartlett's test of sphericity.22 The KMO value of 0.56 and the significant Bartlett's test of sphericity (P< 0.001) in this validation was acceptable. Cronbach's alpha was 0.736, indicating good internal consistency.

Personal details, medical history and contact number of all patients who underwent MAC within the specified period were collected from patient's medical records with the permission from the Head of Breast and Endocrine Unit, Department of General Surgery, HKL. Each patient who fulfilled the selection criteria was assigned a study number and grouped into either conventional analgesic therapy (Group A) or Pecs II block (Group B).

All patients included in this study had undergone MAC under GA with regular method of induction and maintenance inhalational anesthesia. Those who received Pecs II block had the procedure done before induction of anesthesia by a team of experienced regional anesthesiologists. Both groups received appropriate doses of opioid and nonsteroidal anti-inflammatory drugs (NSAID) for intraoperative analgesia. Post operatively, all patients received standardized oral analgesics for pain control.

The survey was conducted by a single investigator. Recruited patients were seen in the surgical outpatient clinic to obtain consent and complete the questionnaire. Patients who were not seen in the clinic were contacted by telephone to obtain verbal consent and answer the questionnaire according to the template prepared (Appendix 2). A series of questions related to chronic pain of PMPS were asked as per questionnaire.

Using Krejcie and Morgan formula,24 sample size was calculated based on the incidence of PMPS, which was our primary outcome variable. Published data showed that the incidence of PMPS ranges from 11% to 60%.7-10 With expected incidence of 60%, using 2 proportions sample test, we calculated that a minimum of 95 patients per study group would provide 80% power (α = 0.05).

Data were analyzed using SPSS version 23.0 software. Continuous variables are presented as mean ± standard deviations or median (interquartile range) where appropriate. Categorical data is shown as numbers and percentages. Comparison of continuous data between groups was performed by Student's

ELIGIBILITY:
Inclusion Criteria:

* patient underwent unilateral mastectomy for breast carcinoma

Exclusion Criteria:

* past history of chronic pain and on regular analgesics, chemotherapy or radiotherapy before surgery, surgical complications (such as infection or wound breakdown) or cancer recurrence, history of psychiatric illness, inability to be contacted, inability or unwillingness to participate in the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient underwent unilateral mastectomy for breast carcinoma
Sampling Method: Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Incidence of PMPS | 2 years
  Incidence of Post mastectomy pain syndrome (PMPS)

SECONDARY OUTCOMES:
Severity of PMPS | 2 years
  Severity of Post mastectomy pain syndrome (PMPS)

CONTACTS AND LOCATIONS:
Overall Officials: YEOH CHIH NIE, Mmed, Principal Investigator — Universiti Kebangsaan Malaysia Medical Centre
Locations (1):
- Universiti Kebangsaan Malaysia Medical Center, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided